CLINICAL TRIAL: NCT05706857
Title: Evaluation of the Clinical Impact of Ultra Fast-Track in Patients Undergoing Cardiac Surgery Versus Conventional Extubation (CARDU-FAST)
Brief Title: Evaluation of the Clinical Impact of Ultra Fast-Track in Patients Undergoing Cardiac Surgery
Acronym: CARDU-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Lourdes Montero Cruces, Cardiovascular Surgeon, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 22/720-EC_X
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Disease; Surgery; Anesthesia
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomized 1:1. Stratified by type of surgery (CABG, Valvular, Aorta)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultra fast-track (Experimental): Patients are extubated in the operating room after the procedure
  Interventions: Behavioral: Ultra Fast-track
- Conventional extubation (Active Comparator): Patients are extubated in the intensive unit care
  Interventions: Behavioral: Ultra Fast-track

INTERVENTIONS:
Behavioral: Ultra Fast-track — Patients are extubated in the operating room

SUMMARY:
Single center randomized clinical trial. The main aim is to demonstrate the superiority at the clinical level of the ultra fast-track programs versus conventional early postoperative extubation in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The study is aimed to compare clinical superiority of ultra fast-track versus conventional early postoperative extubation in patients undergoing cardiac surgery in our center. The estimated sample size is 612 patients. They will be randomized 1:1 to any of the two arms of the study (ultra fast-track vs. fast-track). The randomization will be stratified according the type of surgery performed. The period of recruitment will start in January 2023 and is supposed to finish by September 2024 or earlier. The main outcomes of the study will be measured 1 year after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with valvular, coronary or aortic heart disease with an indication for major cardiac surgery.
* The patient's desire to participate in the clinical trial verified by signing the informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Emergent surgery or cardiorespiratory arrest.
3. Patient in preoperative cardiogenic shock, or in need of high-dose vasoactive support.
4. Aortic arch procedures.
5. Procedures in which hypothermia < 28ºC of temperature is expected during the intervention.
6. Minor cardiac surgery procedures.
7. Procedures with minimally invasive techniques without extracorporeal circulation (Transcatheter aortic valve implantation, Transcatheter mitral valve implantation, Minimally invasive mitral valve repair (TOP-Mini), Totally thoracoscopic MAZE procedure, Minimally invasive direct coronary artery bypass grafting).
8. Implantation of circulatory assistance devices or ECMO (extracorporeal membrane oxygenation).
9. Active endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Determine the effect of Ultra Fast-track | 1 year
  Determine the effect of Ultra Fast-track on the occurrence of the composite outcome composed of all-cause mortality, respiratory complications (prolonged intubation over 24h, reintubation, or pneumonia) and AKIN-III (acute renal failure) in patients undergoing ultra fast-track and patients with conventional postoperative extubation.

SECONDARY OUTCOMES:
Procedural resources conpsumption | 1 year
  Comparison of operating room occupancy time (minutes), ICU stay and overall postoperative stay (days).
Differences in the need for high flow nasal oxygen therapy or non-invasive ventilation for >24h. | 1 year
  Comparison of the need for high flow nasal oxygen therapy or non-invasive ventilation for >24h after the procedure.
Differences in major bleeding or life-threatening bleeding. | 1 year
  Comparison of the event of major bleeding or life-threatening bleeding (VARC 2 definition).
Differences in neurological complication | 1 year
  Comparison of the incidence of neurological complication after the procedure.
Differences in the incidence of acute myocardial infarction. | 1 year
  Comparison of the incidence of acute myocardial infarction after the procedure.
Differences in the incidence of heart reoperation | 1 year
  Comparison of the reoperation rate after the procedure.
Differences in the incidence of infections rate. | 1 year
  Comparison of the incidence of infection that requires intravenous antibiotic therapy, which causes an increase in hospital stay or engage patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Montero Cruces, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain